CLINICAL TRIAL: NCT04057950
Title: Multicentric, Randomized, Double Blind Study Under Dermatological Control for Evaluation of the Antidandruff Maintenance Effect of One Shampoo (Reference 1144628 D) Versus Its Vehicle (Reference 1144781) During 8 Weeks After a Ketoconazole-based Antifungal Treatment During 4 Weeks in Adult Subjects (Male and Female) With Light to Moderate Seborrheic Dermatitis
Brief Title: Effects on the Scalp Microbiota of a 1% Selenium Disulfide and 1% Salicylic Acid Shampoo After 2% Ketaconazole Foaming Gel Treatment for Scalp Seborrheic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 17-00182
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Scalp Dermatitis; Dermatitis
Keywords: seborrheic dermatitis; microbiota; malassezia; bacteria; diversity
MeSH Terms: conditions — Dermatitis; Dermatitis, Seborrheic | interventions — Cosmetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treating shampoo (Active Comparator): treating shampoo (1% Selenium Disulfide (SeS2)/1% salicylic acid-based shampoo) 1144628 D cosmetic product
  Interventions: Other: cosmetic product
- vehicle (Placebo Comparator): 1144781 cosmetic product
  Interventions: Other: cosmetic product

INTERVENTIONS:
Other: cosmetic product — Disulfure de sélénium versus placebo formula
  Other Names: vichy dercos

SUMMARY:
The aim of this study was to investigate the changes in the scalp bacterial and fungal microbiota in subjects afflicted with a scalp seborrheic dermatitis (SSD) during a 2% ketoconazole-based treatment followed by a maintenance phase (1% Selenium Disulfide (SeS2)/1% salicylic acid-based shampoo versus its vehicle).

DETAILED DESCRIPTION:
Seborrheic dermatitis is a chronic, recurrent, cutaneous inflammatory condition that causes erythema and skin flaking, sometimes appearing as macules or plaques with dry white or moist oily scales. In general, this condition affects patients in good general health.

In adults, it commonly occurs in areas with high concentrations of sebaceous glands. The scalp is the most frequently affected area (80-90 percent of the cases).

These plaques are usually masked by the hair but covered by abundant dandruff, very visible on the head and even on the clothes. In the severe forms, the dandruff plaques develop into "helmets": they then cover tufts of hair and can cause them to fall.

On the scalp, the lesions may range from mild desquamation to brownish crusts affixed to the skin and hair. Some patients report pruritus, particularly if the scalp is affected. Secondary bacterial infection may occur, aggravating erythema and exudate and causing local discomfort.

Dandruff is regarded as a mild non-inflammatory form of seborrheic dermatitis. The cause of seborrheic dermatitis is not well understood, but its occurrence appears to be related to the proliferation of commensal Malassezia species.

Seborrheic dermatitis often has a substantial negative impact on quality of life and is associated with direct and indirect medical costs.

The primary goals of therapy for seborrheic dermatitis are to clear the visible signs of disease and reduce bothersome symptoms, especially pruritus. Seborrheic dermatitis of the scalp is most conveniently treated with shampoos containing antifungal agents, corticosteroids, or keratolytic agent. They have been shown to be effective in the treatment of seborrheic dermatitis, but recurrence is common and that ongoing treatment may be necessary.

For this study, the choice of the treatment against seborrheic dermatitis was set to ketoconazole, which is a common treatment that shows efficacy.

The purpose of this study is to find a way to ameliorate the quality of life of subjects with seborrheic dermatitis. This trial will evaluate the antidandruff maintenance effect of a 1% selenium sulfide/1% salicylic acid-based shampoo (cosmetic shampoo) versus its vehicle during a 8 week application duration, after the subjects were treated with a classic antifungal treatment for seborrheic dermatitis (in this study, the treatment will be a ketoconazole-based antifungal treatment for 4 weeks in adults with light to moderate seborrheic dermatitis).

ELIGIBILITY:
Inclusion Criteria:

* Subject with hair length > 2 cm.
* Subject exhibiting a slight to moderate seborrheic dermatitis on the scalp after clinical examination, on D0.
* Subject exhibiting slight to severe squame state of scalp: Total squame score (adherent + non-adherent) ≥ 4 (ranging from 0 to 10) including an adherent squame score ≥ 2.5 (ranging from 0 to 5) and no limit for non-adherent squame score on D0.
* Subject usually using a shampoo 3 times a week and accepting to follow this rate during the whole study period.
* Subject having stopped any possible antidandruff treatment at least 2 weeks prior to D0.
* Subject usually using seborrheic dermatitis treatments

Exclusion Criteria:

* • Main Inclusion Criteria:
* Subject with hair length > 2 cm.
* Subject exhibiting a slight to moderate seborrheic dermatitis on the scalp after clinical examination, on D0.
* Subject exhibiting slight to severe squame state of scalp: Total squame score (adherent + non-adherent) ≥ 4 (ranging from 0 to 10) including an adherent squame score ≥ 2.5 (ranging from 0 to 5) and no limit for non-adherent squame score on D0.
* Subject usually using a shampoo 3 times a week and accepting to follow this rate during the whole study period.
* Subject having stopped any possible antidandruff treatment at least 2 weeks prior to D0.
* Subject usually using seborrheic dermatitis treatments

  • Main Non-Inclusion Criteria:
* Subject who has skin marks on the scalp that could interfere with the assessment (pigmentation trouble, scar elements…).
* Subject who used topic treatment for the scalp (anti-dandruff, anti-hair loss, soothing) or corticosteroid treatment (per os or topical) during the last two weeks before the start of the study.
* Subject with personal history of allergy and/or particular reactivity to antidandruff products.
* Subject with personal history of allergy and/or adverse reactions to cosmetic products containing tensioactive agents
* Subject who has taken: corticoids within 2 weeks before the study entrr, or anti-histaminic, anti-fungal, non-steroidal anti-inflammatory, immunosuppressive, or lithium-based drugs less than 1 month before the study entry, or retinoid acid (local or per os) since less than 6 months before study entry.
* Subject with cutaneous affection of the scalp other than seborrheic dermatitis (psoriasis, alopecia in vertex, pediculosis, atopic dermatitis …).
* Subject affected by serious, non-stabilized or progressive disease as diabetes, hypertension, hypothyroidism or hyperthyroidism which may influence the evolution of studied cutaneous state and morphology.
* Subject affected by serious pathology (cancer, immune-depressed)
* Subject who has undergone a surgical operation in the previous month of the study or having planned it during the study.
* Subject who has started, stopped or changed of hormonal treatment (including contraceptive pill) in the previous 6 weeks.
* Pregnancy or breastfeeding during the last 6 months, ongoing or planned during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Antisquame efficacy of the tested shampoo versus its vehicle with Visual Analog Scale after 8 weeks | before and after 8 weeks of treatement
  Change at 8 weeks versus Baseline at 8 weeks of the squamous scale of the shampoo versus vehicle

SECONDARY OUTCOMES:
Change in scalp microbiome (quantification) | before and after 8 week treatment period.
  change in scalp microbiome (quantification by Polymerase Chain Reaction of Staphylococcus, Propionibacterium, Malassezia)
change in scalp microbiome (qualification) | before and after 8 week treatment period.
  change in scalp microbiome (qualification by Next-Generation Sequencing to evaluate diversities)

CONTACTS AND LOCATIONS:
Overall Officials: Yorik DROUAULT, MD, Principal Investigator — INTERTECK
Locations (1):
- Interteck, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Antidandruff maintenance effect Comparison of the antidandruff maintenance effect, after a 4 weeks treatment with ketoconazole, of two shampoos (active versus vehicle) applied during 8 weeks i.e. up to week 12 (principal objective) and during 4 and 6 weeks i.e. at week 8 and week 10 (secondary objective).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: early 2020